CLINICAL TRIAL: NCT05509439
Title: A Home Transfusion Program for Patients With Advanced Hematologic Malignancies
Brief Title: Home Transfusion for HEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Oreofe Odejide, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-178
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy
Keywords: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Transfusion (Experimental): This research study involves completing questionnaires, a brief interview, blood draws, and blood transfusions when needed.
  * Home Transfusion Program Components
  * Participants will be in the research study for up to six months
  Interventions: Other: Home Transfusion Program Components

INTERVENTIONS:
Other: Home Transfusion Program Components — The Home Transfusion Program will include trained transfusion nurse(s) who will administer transfusions in the home setting. The transfusion nurse, who is part of the study team, will work closely with the DFCI/BWH Blood Bank and the hospice agency (Care Dimensions Inc.) that all study patients are enrolled in. The transfusion nurse will administer home transfusions using safe home transfusion practices endorsed by the AABB. The home transfusion program has 4 key aspects Initial home visit, (2) subsequent contact, (3) home transfusion assessment & administration, (4) usual elements of hospice

SUMMARY:
The purpose of the research is to assess the feasibility and acceptability of a home blood transfusion program for patients with hematologic malignancies who need blood transfusions

DETAILED DESCRIPTION:
This feasibility study will be used to assess the feasibility and acceptability of a hospice-embedded home transfusion program to patients with hematologic malignancies. All enrolled subjects will be patients cared for at Dana Farber Cancer Institute.

This study is a single-arm study of 10 patients with advanced hematologic malignancies who have a limited life-expectancy of six months or fewer and are hospice eligible.

10 Caregivers of enrolled patients will also be invited to participate if interested.

This research study involves completing questionnaires, a brief interview, blood draws, and blood transfusions when needed.

Participants will be in the research study for up to six months.

It is expected that about 20 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced hematologic malignancies:

  * Diagnosis of a hematologic malignancy
  * Age ≥ 18 years
  * Receipt of primary oncologic care at DFCI (at least 2 outpatient visits in 12 months prior to enrollment)
  * Has received at least one red blood cell (RBC) or platelet transfusion since blood cancer diagnosis in the clinic or hospital setting without a serious adverse transfusion reaction
  * Physician-estimated prognosis of six months or less
  * Has an adult informal caregiver that lives in the same residence
  * Patient resides within catchment served by Care Dimensions Hospice
* Caregivers:

  * Identified informal caregiver of enrolled patient with hematologic malignancy
  * Age ≥ 18 years

Exclusion Criteria:

* Patients

  * Age < 18 years
  * Does not have an identified adult informal caregiver who lives in the same residence
  * History of previous serious adverse transfusion reaction
  * Presence of decompensated congestive heart failure
* Caregiver

  * Age < 18 years
  * Our study will exclude members of the following special populations:

    * Adults unable to consent
    * Individuals who are not yet adults (infants, children, teenagers)
    * Pregnant women
    * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Enrollment Rate | 6 months
  Number of patients consented to the study divided by eligible patients approached by the study team
Completion of Home Transfusions and Patient-Reported Data | 6 months
  Proportion of completed home transfusions among enrolled patients who meet transfusion criteria, and proportion of enrolled patients who complete patient-reported data collection

SECONDARY OUTCOMES:
Satisfaction Rate | 3 Weeks
  Proportion of enrolled patients who are satisfied with the home transfusion program and proportion of enrolled patients who are likely to recommend the home transfusion program.
Disenrollment Rate | 6 months
  Proportion of study participants who disenroll from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Oreofe O Odejide, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu